CLINICAL TRIAL: NCT02610673
Title: WiCS-LV Post Market Surveillance Registry
Status: Active, not recruiting | Type: Observational
Sponsor: EBR Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: EBR-02821
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2025-03-21 (Actual); Status verified 2024-07

CONDITIONS: Cardiac Resynchronization Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: WiCS-LV System — Implant of left ventricular receiver-electrode and ultrasound transmitter.
  Other Names: Wireless Cardiac Stimulation; Wireless Stimulation on the Endocardium - WiSE System

SUMMARY:
This is an observational, prospective, non-randomized collection of defined clinical data under normal conditions of use for the WiCS-LV System, an implantable cardiac pacing system capable of delivering pacing energy to the left ventricle of the heart without using a pacing lead.

Patients will be enrolled and followed according to standard of care for 5 years.

DETAILED DESCRIPTION:
A clinical registry will be used to collect data from all implanted patients, at all follow-ups and across all implanting centers. Implant procedure will be according to the 'Instruction for Use' of the system and assessments and follow-ups according the best clinical practice.

Anonymized data will be collected on Case Report Forms (CRF) for each patient in the registry. These data will be collected at the time of implant and at scheduled patient in-clinic follow-ups of 1 week, 3 months, 6 months, and 1, 2,3,4,5 years post implant. Patients entering the registry will be given a Registry code suitable to uniquely identify the patient, the implanting center, and the responsible physician.

Data will be consolidated into a dataset by the sponsor for analysis purposes. The sponsor may request support from the center to review patient records in order to monitor the data in cases where the data appears incomplete or appears to be inaccurate.

The data set will be consolidated such that each implanting center may access its own data, or as mutually agreed between centers, aggregate data. Data may be used by centers for purposes of publication or other objectives of the center.

ELIGIBILITY:
Inclusion Criteria:

Patients with heart failure meeting standard criteria for CRT based upon the current European Society of Cardiology / European Heart Rhythm Association (ESC/EHRA) guidelines and meeting criteria in one of these categorizations:

Untreated by conventional CRT:

This includes:

* Patients that have had an attempted but failed CS lead implant due to such complications as venous occlusion, difficult CS access or anatomy, poor lead stability or previous CS repositioning procedures.
* Patients with a previously implanted CS lead that is programmed off due to such complications as high pacing threshold, non-capture, phrenic nerve stimulation, lead failure, lead dislodgement, or other justifications due to lead issues documented by the prescribing physician.

Non-responder to conventional CRT

This includes:

• Patients with a previously implanted CRT device who based on prescribing physician judgment experience no change or worsening of heart failure symptoms or no change or worsening of NYHA functional class after 6 months of CRT treatment.

Upgrade:

This includes:

* Patients that have a relative contraindication for a CS lead implant such as difficult subclavian access, venous thrombosis, venous occlusion, risk of lead dislodgment, or other justification documented by the prescribing physician.
* Patients that have a relative contraindication for revising an implanted device to a CRT device such as previous pocket erosion, previous pocket infection, previous explantations, or other justifications documented by the prescribing physicians.
* Patients with other justifications based upon the prescribing physician's judgment of risk to reopening the device pocket including consideration for the remaining longevity of the pacemaker/ICD battery.

Exclusion Criteria:

Triple anticoagulation therapy (warfarin, clopidogrel, ASA, or other agents) Stage 4 or 5 renal dysfunction defined as GFR <30 Grade 4 mitral valve regurgitation Thrombocytopenia (platelet count <150,000) Non-ambulatory (or unstable) NYHA class 4 Contraindication to heparin Contraindication to both chronic anticoagulants and antiplatelet agents Contraindication to iodinated contrast agents Insufficient acoustic window to the LV as assessed from diagnostic transthoracic echocardiography Left atrial or left ventricular thrombus Attempted implant of a Pacemaker, ICD, or CRT device within 3 days Life expectancy < 12 months Chronic hemodialysis Myocardial infarction within one month Major cardiac surgery within one month Incompatible electrical stimulation therapy devices, for example transcutaneous electrical nerve stimulation (TENS) or other neurological stimulation devices Exposure to magnetic resonance imaging (MRI) Use of diathermy Use of therapeutic ultrasound Use of echocardiography imaging using vascular, intracardiac, Doppler, and trans-esophageal probes and systems Use of ionizing radiation treatments

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure meeting standard criteria for CRT based upon the current European Society of Cardiology / European Heart Rhythm Association (ESC/EHRA) guidelines and meeting inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-02-08 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Complications | 24 hour perioperative, one month
  Device and procedure related complications
Performance | six months
  Bi-ventricular capture on 12 lead EKG

SECONDARY OUTCOMES:
Device Complications | six months
  Device and procedure related complications
Major Complications | six months
  All major complications
Complications | annually to 5 years
  Device and procedure related complications
Performance | annually to 5 years
  Bi-ventricular capture on 12 lead EKG
Evidence of Efficacy | 6 months
  Clinical composite score (All-cause mortality, HF hospitalizations, NYHA class, and patient global assessment)

CONTACTS AND LOCATIONS:
Locations (3):
- Aalborg University Hospital, Aalborg, Denmark
- Herzzentrum Brandenburg, Bernau, Germany
- Cardiocentro Ticini, Lugano, Switzerland

REFERENCES:
- [Derived] Sieniewicz BJ, Betts TR, James S, Turley A, Butter C, Seifert M, Boersma LVA, Riahi S, Neuzil P, Biffi M, Diemberger I, Vergara P, Arnold M, Keane DT, Defaye P, Deharo JC, Chow A, Schilling R, Behar J, Rinaldi CA. Real-world experience of leadless left ventricular endocardial cardiac resynchronization therapy: A multicenter international registry of the WiSE-CRT pacing system. Heart Rhythm. 2020 Aug;17(8):1291-1297. doi: 10.1016/j.hrthm.2020.03.002. Epub 2020 Mar 9. PMID 32165181